CLINICAL TRIAL: NCT00698568
Title: Study to Evaluate the Safety of GSK Biologicals' Herpes Simplex Candidate Vaccine (gD2t) With MPL in HSV Seropositive or Seronegative Subjects Without Genital Herpes Disease
Brief Title: Safety Evaluation of Herpes Simplex Candidate Vaccine (gD2t) With Adjuvant in HSV Seropositive / Seronegative Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208141/016
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Prophylaxis for Herpes Simplex
Keywords: Herpes simplex, Herpes simplex candidate vaccine
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Herpes simplex candidate vaccine- adjuvanted GSK 208141
- Group B (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes simplex candidate vaccine- adjuvanted GSK 208141 — Intramuscular injection, 3 doses
  Arms: Group A
Biological: Placebo — Intramuscular injection, 3 doses
  Arms: Group B

SUMMARY:
This study will evaluate, versus a placebo, the safety of Herpes simplex candidate vaccine with adjuvant in initially HSV seropositive or seronegative subjects who have no genital herpes disease.

DETAILED DESCRIPTION:
This study was monitored by a Data Safety Monitoring Board. At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over at the time of first vaccination
* Written informed consent
* Females of childbearing potential must have a negative pregnancy test at enrollment and prior to each vaccination and be using an accepted method of birth control

Exclusion Criteria:

* Any previous history of or current clinical signs or symptoms of genital herpes disease.
* Any previous vaccination against herpes simplex.
* Any previous administration of MPL.
* History of herpetic keratitis.
* History of erythema multiforme.
* Female subjects who are pregnant, lactating or planning a pregnancy before one month after the last vaccine dose
* Patient is immuno-compromised or is receiving immuno-modifying therapy of any kind. Topical corticoid therapy is allowed.
* HIV positive at the time of enrollment
* Clinical signs of acute or febrile illness at the time of entry into the study.
* Any continuous suppressive antiviral oral therapy within the 6 months prior to entry.
* Any administration of immunoglobulins during the vaccination course or within one month prior to the first vaccination.
* Any vaccine administration less than one week before or after a study vaccination.
* Previous known hypersensitivity to vaccination or to any component of the vaccine.
* Simultaneous participation in any other clinical trial of an investigational drug or vaccine concurrent with this study or during the period beginning 30 days prior to entry into the study or 5 half-lives of the drug
* Recent history of alcoholism or drug abuse
* Recent clinical history or evidence of significant hepatic disease
* History of a current acute or chronic auto immune disease.
* Recent clinical history or evidence of renal dysfunction
* Life-threatening or serious cardiac (NYHA grades III-IV), gastrointestinal, haematological or immunological disorder which, in the opinion of the investigator, would preclude entry into the study.
* Inability or unwillingness to comply with the protocol or not expected to complete the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7460 (Actual)
Dates: Start 1996-10; Primary Completion 1999-04 (Actual); Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
To compare between herpes simplex vaccine and placebo recipients the general safety of the vaccine by recording all the unsolicited adverse experiences and all serious adverse experiences | During a 30-day period after each vaccination (AEs), during 7 months after study start (SAEs)

SECONDARY OUTCOMES:
To compare between vaccine and placebo recipients the incidence and severity of the reactogenicity as measured by recording the local reactions and the general symptoms | On the day of each vaccination and on the following 3 days
To compare between vaccine and placebo recipients the effect on the haematological and biochemical parameters in subjects from 20% of the centers in each country | At day -90 to day -7, and at month 7 and month 13
To compare between vaccine and placebo recipients the effect on pre-existing herpes simplex virus infection by recording the frequency and severity of all herpes simplex clinical episodes | Day 0 through month 19
To evaluate the incidence and the types of the serious adverse experiences in both groups | Month 7 to month 19
To evaluate the humoral immune response to the vaccine by measuring the anti-gD2 antibodies in a subset of vaccine and placebo recipients from each of the serostatus groups | Before vaccination, and one month and 7 months after vaccination
To compare the anti-gD2 antibody responses between the subsets of HSV double seronegative and HSV-1 seropositive only vaccine recipients | At months 7 and 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (45):
- United States (34):
  - GSK Clinical Trials Call Center, La Jolla, California
  - GSK Clinical Trials Call Center, Middle Valley, California
  - GSK Clinical Trials Call Center, San Diego, California
  - GSK Clinical Trials Call Center, Denver, Colorado
  - GSK Clinical Trials Call Center, East Lyme, Connecticut
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Indianapolis, Indiana
  - GSK Clinical Trials Call Center, Des Moines, Iowa
  - GSK Clinical Trials Call Center, Mission, Kansas
  - GSK Clinical Trials Call Center, Louisville, Kentucky
  - GSK Clinical Trials Call Center, Towson, Maryland
  - GSK Clinical Trials Call Center, Newton, Massachusetts
  - GSK Clinical Trials Call Center, Lansing, Michigan
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Omaha, Nebraska
  - GSK Clinical Trials Call Center, Albuquerque, New Mexico
  - GSK Clinical Trials Call Center, Brooklyn, New York
  - GSK Clinical Trials Call Center, Poughkeepsie, New York
  - GSK Clinical Trials Call Center, Cincinnati, Ohio
  - GSK Clinical Trials Call Center, Portland, Oregon
  - GSK Clinical Trials Call Center, Philadelphia, Pennsylvania
  - GSK Clinical Trials Call Center, Pittsburgh, Pennsylvania
  - GSK Clinical Trials Call Center, Providence, Rhode Island
  - GSK Clinical Trials Call Center, Charleston, South Carolina
  - GSK Clinical Trials Call Center, Austin, Texas
  - GSK Clinical Trials Call Center, Bryan, Texas
  - GSK Clinical Trials Call Center, Dallas, Texas
  - GSK Clinical Trials Call Center, Lake Jackson, Texas
  - GSK Clinical Trials Call Center, Nassau Bay, Texas
  - GSK Clinical Trials Call Center, San Antonio, Texas
  - GSK Clinical Trials Call Center, Salt Lake City, Utah
  - GSK Clinical Trials Call Center, Falls Church, Virginia
  - GSK Clinical Trials Call Center, Seattle, Washington
  - GSK Clinical Trials Call Center, Wenatchee, Washington
- GSK Clinical Trials Call Center, Sydney, New South Wales, Australia
- GSK Clinical Trials Call Center, Vienna, Austria
- GSK Clinical Trials Call Center, Ghent, Belgium
- GSK Clinical Trials Call Center, Montreal, Quebec, Canada
- GSK Clinical Trials Call Center, Copenhagen, Denmark
- GSK Clinical Trials Call Center, Grenoble, France
- GSK Clinical Trials Call Center, München, Germany
- GSK Clinical Trials Call Center, Carolina, Puerto Rico
- GSK Clinical Trials Call Center, Pretoria, South Africa
- GSK Clinical Trials Call Center, Madrid, Spain
- GSK Clinical Trials Call Center, Basel, Switzerland